CLINICAL TRIAL: NCT01314521
Title: Suicidal Ideation and Behavior in Korean Adolescents With Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Collaborators: Bundang CHA Hospital (Other); Myongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SKAD
Record Dates: First submitted 2011-03-09; First posted 2011-03-14 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-03

CONDITIONS: Depression
Keywords: Suicide; Depression; Adolescents
MeSH Terms: conditions — Depression; Suicide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to examine clinical characteristics of Korean adolescents with depression who have suicidal ideation and behavior. We formulate those hypotheses.

1. Being bullied in peer relationships, excessive use of internet, excessive extra-curricular tutoring, sexual abuse in childhood, physical abuse and emotional neglect are risk factors of suicide in adolescents.
2. Depression of parents and negative child-rearing attitude are risk factors of suicidal ideation and behavior in adolescents.
3. Emotional quotient (EQ) and resilience of adolescent are protective factors of suicide.

DETAILED DESCRIPTION:
Korea has reported the highest suicide rate among OECD members and according to the data from the Korea national statistical office, suicide is the second major cause of death in adolescents and is increasing. Depression, one of the well-known risk factors of suicide in adolescents, can cause maladjustments to school and family life, problems of interpersonal relationship and drug abuse so that work to trigger the suicidal ideation and behavior. In his study, we planned to examine the relationship between suicidal ideation and behavior and several risk factors by using the standardized diagnostic clinical interview, especially an objective suicide evaluating method which has recently developed.

ELIGIBILITY:
Inclusion Criteria:

* a subject who has depression (Major depressive disorder, dysthymic disorder, depressive disorder NOS) diagnosed by Kiddie-Schedule for affective disorder and schizophrenia (K-SADS-PL-K)
* subjects and their family (a parent or a grandparent) or their legal representative consent to participate in this study voluntarily
* subjects and their family (a parent or a grandparent) or their legal representative are able to understand the meaning of participation in this study and able to reject or ask to leave from this study

Exclusion Criteria:

* a patient who has diagnosed with bipolar disorder, psychotic disorder, pervasive developmental disorder, organic brain disease, or epilepsy
* a patient with mental retardation who is IQ under 70
* a patient who has a severe medical illness (chronic physical disease, cardiovascular, hepatobiliary, nephrology, or respiratory disease and so on)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: outpatients of university hospitals. 50 from Hallym University Sacred Heart Hospital, 50 from Bundang CHA Hospital, 50 from Myongji Hospital.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-01; Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Columbia Suicide Severity Rating Scale; C-SSRS | baseline only (at any one point during the depressive episode)
  Semi-structured clinical interview based on the systematic guideline which help draw inferences about suicidal ideation from clinical situation and risk factors related to the suicide. It is composed with three categories that are suicidal attempt (ideation), non-suicidal attempt (ideation), and potential of suicidal attempt (ideation).

SECONDARY OUTCOMES:
Beck suicidal ideation scale | baseline only
  self report form of 19 items with 3 point scale. for subjects and their parents.
Revised Children's Manifest Anxiety Scale; RCMAS | baseline only
Beck Depression Inventory | baseline only

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Ju Hong, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Kyeonggi Do, South Korea